CLINICAL TRIAL: NCT05375175
Title: Estudio de Las Propiedades Saciantes de un Snack de proteína híbrida Proveniente Mayoritariamente de Garbanzos
Brief Title: Study of the Satiating Properties of a Hybrid Protein Snack Mainly From Chickpeas
Acronym: LegumSnacks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IDI-20190984
Record Dates: First submitted 2022-04-20; First posted 2022-05-16 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-04

CONDITIONS: Healthy Nutrition

STUDY DESIGN:
Intervention Model Description: A randomized, crossover and controlled clinical trial will be developed with 23 individuals to evaluate the post-prandial effect of consuming snacks rich in vegetable and animal protein compared to a high-quality pork sausage. Each participant will consume the 2 types of snacks (20 grams) following a random assignment order.
  It is a randomized, crossover, double-blind, and controlled trial. The intervention will consist of the administration of 20 g of one or another snack (Fertinagro Company) that will be eaten at fasting in the morning. Participants will be fasting for 12 hours for solid or liquid food and more than 1 hour after ingestion of water. Blood samples will be obtained after venepuncture at 7:45 a.m. before eating snacks and 15, 30, 60, 90 and 120 minutes after it.
  Within a period of 20 days +_5 days, the intervention will be carried out with the second type of snack according to randomization. The total duration of the study is expected to be 2.5 to 3 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To ensure double-blindness, the wrapper of the snacks will be the same and nursing will only be able to distinguish the product by the assigned code, as will the statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Snack (Experimental): Hybrid Snack: combination of legumes, in the highest proportion, and lean meat.
  Interventions: Other: Hybrid Snack
- Meat snack (Active Comparator): Meat snack: composed of meat from loin tape
  Interventions: Other: Meat snack

INTERVENTIONS:
Other: Hybrid Snack — The intervention will consist of the administration of 20 g of the snack (produced by Fertinagro Company) that will be eaten at fasting in the morning. Participants will be fasting for 12 hours for solid or liquid food and more than 1 hour after ingestion of water. Blood samples will be obtained after venepuncture at 7:45 a.m. before eating snacks and 15, 30, 60, 90 and 120 minutes after it.
  Hybrid snack: combination of legumes in the highest proportion and lean meat.
  It will have the following composition:
  Ingredients (%):
  Chickpea flour 45.40% Natural emulsifier 0.40% Meat 15.50% Olive oil 1.00% Sunflower oil 4.00% Water 22.50% Onion powder 0.30% Garlic powder 0.20% Thyme 0.60% Tomato powder 10.00%
  Arms: Hybrid Snack
Other: Meat snack — The intervention will consist of the administration of 20 g of the snack (produced by Fertinagro Company) that will be eaten at fasting in the morning. Participants will be fasting for 12 hours for solid or liquid food and more than 1 hour after ingestion of water. Blood samples will be obtained after venepuncture at 7:45 a.m. before eating snacks and 15, 30, 60, 90 and 120 minutes after it.
  Snack sausage:
  Composed solely of meat from loin tape
  It will have the following composition:
  Ingredients (%):
  Shoulder meat 4 mm 94.13% Low sodium salt 3.30% Maltodextrin 1.65% Spices 0.28% Natural dye 0.64%
  Arms: Meat snack

SUMMARY:
A randomized, crossover and controlled clinical trial will be developed in 23 individuals to evaluate the postprandial effect of consuming snacks rich in vegetable and animal protein compared to a high-quality pork sausage

DETAILED DESCRIPTION:
A randomized, crossover and controlled clinical trial will be developed in 23 individuals to evaluate the postprandial effect of consuming snacks rich in vegetable and animal protein compared to a high-quality pork sausage. Each of the participants will consume the two types of snacks (20 grams) following a random assignment order. The design is randomised and cross-over.

A greater satiating effect is expected with the hybrid snack, given that the fiber in chickpea flour is higher than that of dry chickpeas. In addition, chickpea flour is rich in soluble fiber (a type of fiber that helps retain water and therefore slows down digestion) having positive effects on the gastrointestinal tract and on the metabolism of LDL cholesterol, as well as on blood glucose .

Foods high in complex carbohydrates and fiber have a satiating effect due to their fiber content. It is known that the most satiating macronutrient is protein if the food also contains fiber, this favors that some nutrients are not fully absorbed, including fat. Hence, these foods have a satiety index greater than fat itself, thus favoring adherence to diet and body weight, since it is possible to control portions, avoiding snacking on unhealthy products.

ELIGIBILITY:
Inclusion Criteria:

* 23 participants between 18 and 30 years old, with a ratio between men and women of approximately 50%.

Exclusion Criteria:

* Diabetics
* Chronic medication except contraceptives
* Diagnosis of inflammatory bowel disease (IBD)
* Any serious active disease that prevents or disables to adequately follow the study
* Regular cannabis users
* Alcoholism or active drug dependence
* Inability to give informed consent
* Pregnancy and lactation
* Intolerance to any of the components of the two snack which are intended to be tested

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 23 participants between 18 and 30 years old, with a ratio between men and women of approximately 50% will be recruited
Enrollment: 23 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Satiety | post-prandial state: we will study blood samples before eating snacks and the change at 15, 30, 60, 90 and 120 minutes after it.
  Satiety will be measured through the objective determination of endocannabinoid compounds by mass spectrometer analysis

CONTACTS AND LOCATIONS:
Overall Officials: Montse Fitó, Principal Investigator — Parc de Salut Mar
Locations (1):
- IMIM, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
A consortium agreement will be established with the collaborating partners at the beginning of the project, focusing on confidentiality issues, agreements of all parties and patent possibilities.
  The study data must be verifiable with the source data, which necessitates access to all original records, laboratory reports, and subject records. The confidentiality of the data and the identity of the patients will be maintained during the study and after its completion. Only the Principal Investigator and authorized study personnel will have access to these confidential records.
  The data and other information related to the project is managed through REDCap, a secure web application that is installed on a server located in CIBER. The IP is the repository owner of the information contained in the project database.
  No data used in the analysis and subsequent disclosure of the study results will contain any identifiable reference to patient names.